CLINICAL TRIAL: NCT05809388
Title: Implementation of Parent Training Through the Use of Virtual Reality: a Randomized, Controlled, Single-blind Study
Brief Title: Virtual Reality for Parent Training Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Adriana Piccolo, Principal Investigator, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PT22
Record Dates: First submitted 2023-03-17; First posted 2023-04-12 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Attention-Deficit/Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (EG) (Experimental): The EG will perform a standard Parent Training program. This PT will be supplemented with virtual reality sessions. Each pair of parents will perform a total of 12 treatment sessions fortnightly.
  Interventions: Behavioral: Parent training; Behavioral: Virtual Reality-assisted PT sessions
- Control Group (CG) (Active Comparator): The CG will perform a standard Parent Training program plus two follow up sessions. Each pair of parents will perform a total of 12 treatment sessions fortnightly.
  Interventions: Behavioral: Parent training

INTERVENTIONS:
Behavioral: Parent training — Parent Training program according to "Ten steps of Barkley's program" plus two additional follow-up sessions. This will be conducted by a trained psychologist; each session will last approximately 60 minutes and will includes exercises, discussions and role-playing.
Behavioral: Virtual Reality-assisted PT sessions — The experimental group will follow the same program of CG sample. Parent Training sessions will be conducted by a trained psychologist; each session will last approximately 60 minutes that include:
  * 40 minutes of as usual PT session, with exercises, discussions and role-playing.
  * 20 minutes of VR screen with which the parents may interact; VR screen will provides instructive, stimulating, interactive, and direct feedbacks exercises to enhance parenting strategies.
  Arms: Experimental Group (EG)

SUMMARY:
Previous research has shown how parental responses can affect ADHD symptoms by triggering dysfunctional cyclic processes. Therefore, it may be useful within rehabilitative treatments to include parent training (PT). Recent literature data have demonstrated the potential of using virtual reality in the rehabilitation of children with ADHD. No study has been conducted on the use of virtual reality (VS) within a PT program. It is possible to hypothesize that virtual reality, by providing a controlled environment can help the parent improve his or her ability to self-control and perceive the child's difficulties. This allows the parent's empathizing skills to be implemented and reinforces the educational techniques learned during the parent training intervention.

DETAILED DESCRIPTION:
The investigators designed a single-blind, randomized, controlled study on ADHD patients and their parents, with the aim of evaluating the effects of virtual reality support during PT program compared to traditional PT sessions.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ADHD, according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria;
* Age including 6 to 10 years;
* Subjects with IQ >70;
* Signed informed consent and the availability of at least one family member to participate in the diagnostic/therapeutic process.

Exclusion Criteria:

* Important comorbidities with psychiatric or neurological syndromes (e.g., epilepsy, known genetic syndromes, infantile cerebral palsy, sensory deficits);
* Subjects under the age of 6 years;
* Subjects older than 10 years of age;
* Subjects diagnosed with intellectual disability (IQ ≤70);
* Informed consent not signed and/or unavailability of at least one family member to participate in the diagnostic/therapeutic process.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Parenting Stress Index | Baseline
  Parenting Stress Index is for the early identification of characteristics that may impair normal child development, such as emotional and behavioral disorders and parents who are at risk of living dysfunctionally in their role; Parenting Stress Index has 36 items based on a five-point Likert scale where each value corresponds to a specific statement (1 = completely disagree; 5 = completely agree). The subscale scores range from 12 to 60, and the Total Stress score ranges from 36 to 180. The higher the score, the greater the level of parental stress.
Parenting Stress Index | Month 6
  Parenting Stress Index is for the early identification of characteristics that may impair normal child development, such as emotional and behavioral disorders and parents who are at risk of living dysfunctionally in their role; Parenting Stress Index has 36 items based on a five-point Likert scale where each value corresponds to a specific statement (1 = completely disagree; 5 = completely agree). The subscale scores range from 12 to 60, and the Total Stress score ranges from 36 to 180. The higher the score, the greater the level of parental stress.
Parenting Stress Index | Month 9
  Parenting Stress Index is for the early identification of characteristics that may impair normal child development, such as emotional and behavioral disorders and parents who are at risk of living dysfunctionally in their role; Parenting Stress Index has 36 items based on a five-point Likert scale where each value corresponds to a specific statement (1 = completely disagree; 5 = completely agree). The subscale scores range from 12 to 60, and the Total Stress score ranges from 36 to 180. The higher the score, the greater the level of parental stress.
The World Health Organization Quality of Life | Baseline
  World Health Organization Quality of Life-BREF consists of 26 questions. World Health Organization Quality of Life has Likert-type scoring ranging from 1 to 5. As the score obtained from the sub-domains of the scale increases, the quality of life increases.
The World Health Organization Quality of Life | Month 6
  World Health Organization Quality of Life-BREF consists of 26 questions. World Health Organization Quality of Life-BREF has Likert-type scoring ranging from 1 to 5. As the score obtained from the sub-domains of the scale increases, the quality of life increases.
The World Health Organization Quality of Life | Month 9
  World Health Organization Quality of Life-BREF consists of 26 questions. World Health Organization Quality of Life-BREF has Likert-type scoring ranging from 1 to 5. As the score obtained from the sub-domains of the scale increases, the quality of life increases.
Conners Rating Scale | Baseline
  Conners: a questionnaire that asks about things like behavior, work or schoolwork, and social life. The Conners-3 Parent Rating Scale (Conners-3-P) is the most recent revision to a widely used behavior rating scale system. The Conners-3-P includes 5 empirically derived scales: Hyperactivity/Impulsivity, Executive Functioning, Learning Problems, Aggression, and Peer Relations.Respondents are asked to rate behavior that has been problematic over the preceding month using a four-point Likert scale labeled with both levels of appropriateness (e.g., "Not true at all" = 0), and frequency (e.g., "Very frequent" = 3).
Conners Rating Scale | Month 6
  Conners: a questionnaire that asks about things like behavior, work or schoolwork, and social life. The Conners-3 Parent Rating Scale (Conners-3-P) is the most recent revision to a widely used behavior rating scale system. The Conners-3-P includes 5 empirically derived scales: Hyperactivity/Impulsivity, Executive Functioning, Learning Problems, Aggression, and Peer Relations.Respondents are asked to rate behavior that has been problematic over the preceding month using a four-point Likert scale labeled with both levels of appropriateness (e.g., "Not true at all" = 0), and frequency (e.g., "Very frequent" = 3).
Conners Rating Scale | Month 9
  Conners: a questionnaire that asks about things like behavior, work or schoolwork, and social life. The Conners-3 Parent Rating Scale (Conners-3-P) is the most recent revision to a widely used behavior rating scale system. The Conners-3-P includes 5 empirically derived scales: Hyperactivity/Impulsivity, Executive Functioning, Learning Problems, Aggression, and Peer Relations.Respondents are asked to rate behavior that has been problematic over the preceding month using a four-point Likert scale labeled with both levels of appropriateness (e.g., "Not true at all" = 0), and frequency (e.g., "Very frequent" = 3).

SECONDARY OUTCOMES:
Tower of London Test | T0 (BASELINE) - T1 (SIX MONTHS) - T2 (NINE MONTHS)
  Tower of London Test : is used to assess executive functions, particularly the future implications of one's action
Nepsy- II | T0 (BASELINE) - T1 (SIX MONTHS) - T2 (NINE MONTHS)
  Nepsy battery assess a whole range of general attentional and executive functions, such as the ability to inhibit learned automatic responses, to monitor and self-regulate one's own behaviors and responses, selective and sustained attention (vigilance), the ability to understand, generate, maintain, or change a set of response rules, non-verbal problem-solving skills, and the ability to plan and organize complex responses
Parenting Styles Questionnaire | T0 (BASELINE) - T1 (SIX MONTHS) - T2 (NINE MONTHS)
  This questionnaire assesses the types of parental styles by presenting a list of qualities and behaviors referred to situations of interaction with the child. Answers are collected using a Likert-scale 5-point, from never (=1) to always (=5). Parenting style is measured by calculating as an average over the items related to each style.
Child behavior Checklist | T0 (BASELINE) - T1 (SIX MONTHS) - T2 (NINE MONTHS)
  Child behavior Checklist assesses emotional and behavioral problems in children
Test of Multidimensional self-esteem | T0 (BASELINE) - T1 (SIX MONTHS) - T2 (NINE MONTHS)
  TMA is gets an accurate measurement of self-esteem in developmental age a 150-items self-report questionnaire. It's made up of six subscales: interpersonal relationships, environmental control competence, emotionality, scholastic success, family life, body perception. Participants have to express their agreement with each item according to the following response options: absolutely true, true, false, absolutely false.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Centro Neurolesi Bonino Pulejo, Messina, Italy

REFERENCES:
- [Background] Felt BT, Biermann B, Christner JG, Kochhar P, Harrison RV. Diagnosis and management of ADHD in children. Am Fam Physician. 2014 Oct 1;90(7):456-64. PMID 25369623
- [Background] Lange KW, Reichl S, Lange KM, Tucha L, Tucha O. The history of attention deficit hyperactivity disorder. Atten Defic Hyperact Disord. 2010 Dec;2(4):241-55. doi: 10.1007/s12402-010-0045-8. Epub 2010 Nov 30. PMID 21258430
- [Background] Mulligan A, Anney R, Butler L, O'Regan M, Richardson T, Tulewicz EM, Fitzgerald M, Gill M. Home environment: association with hyperactivity/impulsivity in children with ADHD and their non-ADHD siblings. Child Care Health Dev. 2013 Mar;39(2):202-12. doi: 10.1111/j.1365-2214.2011.01345.x. Epub 2011 Dec 14. PMID 22168816
- [Background] Hosainzadeh Maleki Z, Mashhadi A, Soltanifar A, Moharreri F, Ghanaei Ghamanabad A. Barkley's Parent Training Program, Working Memory Training and their Combination for Children with ADHD: Attention Deficit Hyperactivity Disorder. Iran J Psychiatry. 2014 Apr;9(2):47-54. PMID 25632280
- [Background] Mulvihill A, Carroll A, Dux PE, Matthews N. Self-directed speech and self-regulation in childhood neurodevelopmental disorders: Current findings and future directions. Dev Psychopathol. 2020 Feb;32(1):205-217. doi: 10.1017/S0954579418001670. PMID 30704545
- [Background] Modesto-Lowe V, Danforth JS, Brooks D. ADHD: does parenting style matter? Clin Pediatr (Phila). 2008 Nov;47(9):865-72. doi: 10.1177/0009922808319963. Epub 2008 Jun 16. PMID 18559885
- [Background] Sibley MH, Graziano PA, Ortiz M, Rodriguez L, Coxe S. Academic impairment among high school students with ADHD: The role of motivation and goal-directed executive functions. J Sch Psychol. 2019 Dec;77:67-76. doi: 10.1016/j.jsp.2019.10.005. Epub 2019 Nov 22. PMID 31837729
- [Background] Zwi M, Jones H, Thorgaard C, York A, Dennis JA. Parent training interventions for Attention Deficit Hyperactivity Disorder (ADHD) in children aged 5 to 18 years. Cochrane Database Syst Rev. 2011 Dec 7;2011(12):CD003018. doi: 10.1002/14651858.CD003018.pub3. PMID 22161373
- [Background] Bashiri A, Ghazisaeedi M, Shahmoradi L. The opportunities of virtual reality in the rehabilitation of children with attention deficit hyperactivity disorder: a literature review. Korean J Pediatr. 2017 Nov;60(11):337-343. doi: 10.3345/kjp.2017.60.11.337. Epub 2017 Nov 27. PMID 29234356
- [Background] Venuti, P., & Senese, V. P. (2007). Un questionario di autovalutazione degli stili parentali: Uno studio su un campione Italiano [A questionnaire of self parental styles: A study of an Italian sample]. Giornale Italiano di Psicologia, 34(3), 677-697.